CLINICAL TRIAL: NCT06569758
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Subcutaneous Doses of GenSci098 in TED Patients
Brief Title: A Study of GenSci098 in Subjects With Active Thyroid Eye Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GenSci098-101
Record Dates: First submitted 2024-08-14; First posted 2024-08-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Safety; Tolerability; GenSci098; Thyroid Eye Disease (TED)
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GenSci098 (Experimental)
  Interventions: Drug: GenSci098
- GenSci098 Placebo (Placebo Comparator)
  Interventions: Drug: GenSci098 Placebo

INTERVENTIONS:
Drug: GenSci098 — subcutaneous , 5 dose levels(15mg, 45mg, 90mg, 180mg and 270mg) will be assigned.
  Arms: GenSci098
Drug: GenSci098 Placebo — In SAD part only one dose of GenSci098 and GenSci098 Placebo to be given, in MAD part, multiple doses of GenSci098 and GenSci098 Placebo will be given.
  Arms: GenSci098 Placebo

SUMMARY:
To evaluate the safety and tolerability of single and multiple ascending subcutaneous doses of GenSci098 in patients with thyroid eye disease (TED)

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of single and multiple ascending subcutaneous doses of GenSci098 in patients with thyroid eye disease (TED)

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the informed consent form (ICF): aged between 18 and 75 years (inclusive).
2. Diagnosed by the physician as having active TED associated with Graves' disease (GD), based on clinical and laboratory test results, with a CAS ≥ 3 (on the 7-point scale) for the most severely affected eye at screening and baseline.
3. Onset of active symptoms and signs of TED (including one or more of the following: redness of conjunctiva, swelling of conjunctiva (chemosis), redness of eyelids, swelling of eyelids, swelling of caruncle or plica, spontaneous retrobulbar pain, and pain on attempted upward or downward gaze) within 12 months prior to the screening visit.
4. Positive for thyroid stimulating hormone receptor antibodies (TRAb) at screening.
5. Moderate to severe TED (impacting the quality of life, requiring intervention but not threatening vision), usually with at least 2 of the following manifestations: (1) eyelid retraction width ≥ 2 mm, (2) moderate or severe soft tissue involvement, (3) proptosis ≥ 3 mm above normal for race and gender, (4) inconstant or constant diplopia.
6. Participants must be euthyroid with the underlying disease under control, or have mild hypo- or hyperthyroidism at screening. (Only applicable to Part 1)
7. Participants must have normal thyroid function or hyperthyroidism due to GD at screening. (Only applicable to Part 2)
8. No prior treatment with antithyroid medications and/or thyroid hormone replacement therapy, or having taken antithyroid medications and/or thyroid hormone replacement therapy on a stable dose, or having not been treated with antithyroid medications and/or thyroid hormone replacement therapy due to intolerable side effects.
9. Anyone who will not be required to need or receive any immediate or planned surgical ophthalmological intervention, corrective surgery or orbital irradiation during the study.
10. Female participants must meet one of the following conditions to be eligible for the study:

    1. Infertile, defined as surgical sterilization (hysterectomy, bilateral salpingectomy, bilateral tubal ligation, or bilateral oophorectomy) at least 6 weeks prior to administration or menopausal (spontaneous amenorrhea ≥ 12 months which is not caused by underlying diseases and confirmed by serum follicle stimulating hormone [FSH] level ≥ 40 mIU/mL).
    2. Fertile female participants agree, from the start of the screening visit until 300 day after the last dose, to consistently and correctly use one of the following acceptable methods of effective contraception:

       1. Complete abstinence (based on the participant's preference and usual lifestyle).
       2. Use of oral contraceptives (estrogen and progesterone), and being on a stable dose of the same contraceptive medication for at least 3 months prior to study treatment.
       3. Injectable or implantable hormonal contraception, or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception with similar efficacy (failure rate < 1%), such as a hormonal vaginal ring or transdermal hormonal contraception. 4) Vasectomized partner, with the procedure performed at least 6 months ago.
11. Male participants must meet one of the following criteria to be eligible for the study:

1) agree to use a condom plus an effective method of contraception (i.e., hormonal contraception initiated at least 30 days prior to administration; or placement of an IUD or IUS) when engaging in sexual activity with a female partner of childbearing potential from the start of the screening visit until 24 weeks after the last dose and refrain from donating sperm during this period.

2) agree to practice abstinence from the start of the screening visit until 24 weeks after the last dose.

3) have had a vasectomy at least 6 months prior to study treatment. 12. Voluntarily sign the ICF and be able to understand and comply with the study's treatment regimen and assessments until the end of the study

Exclusion Criteria:

1. Decreased best corrected visual acuity due to optic neuropathy as defined by a decrease in vision of 2 or more lines on the Snellen chart or standard logarithmic chart, new visual field defect, or color defect secondary to optic nerve involvement within the last 6 months.
2. Corneal injury not relieved by medical management.
3. Improvement in CAS of ≥ 2 points within 1 month prior to screening or between screening and baseline.
4. Decrease in proptosis of ≥ 2 mm within 1 month prior to screening or between screening and baseline.
5. Previous orbital irradiation or surgery for TED.
6. Use of any steroid (either intravenous or oral) with a cumulative dose equivalent to ≥ 1 g of methylprednisolone for TED within 4 weeks prior to screening (discontinued steroid eye drops arepermitted).
7. Use of steroids for conditions other than TED within 4 weeks prior to screening (topical steroids for dermatological conditions and inhaled steroids are permitted).
8. Drug therapy with biologics or peptides, including teprotumumab, rituximab, or tocilizumab, within 6 months or 5 half-lives of the drug (whichever is longer) prior to screening.
9. Use of any non-steroidal immunosuppressive agents within the 3 months prior to screening.
10. Pre-existing ophthalmic disease or autoimmune disease (other than TED) that, in the judgment of the investigator, would preclude study participation or complicate interpretation of study results.
11. History of hyperthyroidism not caused by GD (e.g., toxic adenoma or toxic multinodular goiter), and/or current or previous history of thyroid storm. (Only applicable to Part 2)
12. History of radioiodine treatment or thyroidectomy within 6 months prior to first dose. (Only applicable to Part 2)
13. Individuals who cannot abstain from smoking/tobacco products from the screening period to the end of the study.
14. Any known allergy to the components of the investigational product or analogues or previous allergic reactions to monoclonal antibodies.
15. Known history /diagnosis of malignancy.
16. Acute/chronic infection within 2 weeks prior to screening.
17. Participation in another clinical trial within 3 months before screening (except those who did not receive any intervention), or within 5 half-lives of the study drug in other clinical trials (whichever is longer), or concurrent enrollment in another clinical trial.
18. Those with prolonged QTcF interval in 12-lead ECG results (> 450 ms for males, > 460 ms for females) or clinically significant abnormalities in other 12-lead ECG parameters at screening that, in the investigator's judgment, may affect trial participation;
19. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 3 times the ULN, or total bilirubin (TBIL) or alkaline phosphatase (ALP) > 2 × ULN, blood creatinine (Cr) ≥ 1.5 times the ULN at screening.
20. Positive blood pregnancy test, or lactating women at the time of screening.
21. Positive for hepatitis C virus antibody (HCV Ab), human immunodeficiency virus antibody (HIV Ab), Treponema pallidum particle agglutination (TPPA) test, or hepatitis B surface antigen (HbsAg) at screening.
22. History of recreational drug use or substance abuse or positive drug screening results at screening.
23. Any medical (including other clinically significant abnormal laboratory test parameters) or other conditions that the investigator believes might affect the conduct of the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2027-09-02 (Estimated); Study Completion 2027-12-13 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) (physical examination, vital signs, laboratory tests, 12-lead electrocardiogram [ECG]). | SAD Part: 169 days, MAD Part: 281 days

SECONDARY OUTCOMES:
PK parameters after single and multiple subcutaneous doses of GenSci098: maximum concentration at steady state (Cmax,ss); | SAD Part: 169 days, MAD Part: 281 days
PK parameters after single and multiple subcutaneous doses of GenSci098: minimum concentration at steady state (Cmin,ss); | SAD Part: 169 days, MAD Part: 281 days
PK parameters after single and multiple subcutaneous doses of GenSci098: time to maximum concentration at steady state (Tmax,ss); | SAD Part: 169 days, MAD Part: 281 days
PK parameters after single and multiple subcutaneous doses of GenSci098: average concentration at steady state (Cav,ss); | SAD Part: 169 days, MAD Part: 281 days
PK parameters after single and multiple subcutaneous doses of GenSci098: area under the concentration-time curve at steady state (AUC0-τ,ss); | SAD Part: 169 days, MAD Part: 281 days
PK parameters after single and multiple subcutaneous doses of GenSci098: apparent clearance CL/F | SAD Part: 169 days, MAD Part: 281 days
PK parameters after single and multiple subcutaneous doses of GenSci098: half life t1/2, | SAD Part: 169 days, MAD Part: 281 days
Incidences of anti-drug antibodies (ADAs) and neutralizing antibodies (NAbs), and titer of ADA. | SAD Part: 169 days, MAD Part: 281 days

OTHER OUTCOMES:
Changes from baseline in serum inflammatory cytokines including interleukin (IL)-6 | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including interleukin IL-8, | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including monocyte chemotactic protein 1 (MCP-1) | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including interleukin IL-4 | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including interleukin IL-10 | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including interleukin IL-12 | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including interleukin IL-13 | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including interleukin IL-17 | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including interleukin IL-23 | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including interleukin IL-1β | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including soluble interleukin-1 receptor antagonist (sIL-1RA) | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including interferon γ (IFN γ) | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including transforming growth factor β (TGF β) | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including tumor necrosis factor α (TNF α) | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including Chemokine(C-X-C Motif) | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum inflammatory cytokines including Ligand 10 (CXCL-10 | SAD Part: 169 days, MAD Part: 281 days
Change from Baseline in proptosis of the study eye，amount of protrusion of the eye from the orbital rim measured by Hertel exophthalmometer. | SAD Part: 169 days, MAD Part: 281 days
Change from Baseline in CAS value of the study eye,composed spontaneous retrobulbar pain, pain on attempted upward or downward gaze,redness of eyelids,redness of conjunctiva,swelling of caruncle or plica,swelling of eyelids,swelling of conjunctiva. | SAD Part: 169 days, MAD Part: 281 days
Change from Baseline in diplopia，Diplopia assessment will be performed using the Gorman score | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in GO-QoL. | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum thyrotropin receptor antibody (TRAb), | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in thyroid-stimulating antibody (TSAb) | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum total triiodothyronine (T3) | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum total thyroxine (T4) | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum free triiodothyronine (FT3) | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum free thyroxine (FT4) | SAD Part: 169 days, MAD Part: 281 days
Changes from baseline in serum thyroid-stimulating hormone (TSH) | SAD Part: 169 days, MAD Part: 281 days

CONTACTS AND LOCATIONS:
Overall Officials: Huifang Zhou, PHD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's hospital, Shanghai Jiaotong University School of Medication, Shanghai, Shanghai Municipality, China